CLINICAL TRIAL: NCT05746065
Title: A Cohort for Evaluation of Open-label PrEP Delivery and PrEP Preferences Among African Women
Brief Title: A Cohort for Evaluation of Open-label PrEP Use and PreP Preferences Among African Women
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor: School of Medicine, University of Washington
Other Study IDs: STUDY00015634
Record Dates: First submitted 2023-01-05; First posted 2023-02-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine collection to test for syphilis, trichomonas, gonorrhea, chlamydia and HIV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: PrEP — Eligible women will be prescribed PrEP intake in accordance to standard of care should they choose. We are interested in observing adherence, barriers to adherence, and other factors that effect sexual health.
  Other Names: Truvada

SUMMARY:
INSIGHT is a Prospective, Observational, open-label cohort study on women in Sub-Saharan Africa on PrEP screening, informed choice, and compliance.

There are no specific intervention arms or comparative treatment plans. We will follow and observe participants taking PrEP, not taking PrEP, as well as those who begin or end PrEP during the course of the observational period.

DETAILED DESCRIPTION:
Primary goals:

* Estimate HIV incidence using recency testing on samples from women who screen out due to HIV infection, as well as assess HIV incidence prospectively in the cohort.
* Assess the characteristics of women who initiate PrEP compared to those who do not initiate PrEP.
* Evaluate young women's preferences for attributes of long-acting formulations of PrEP, using a discrete choice experiment.
* Assess the acceptability of a patient-facing PrEP decision support tool to provide young women more informed choice about PrEP options.

ELIGIBILITY:
Inclusion Criteria:

* 16-30 years of age
* Female

Exclusion Criteria:

* not sexually active
* over 31 years of age at consent

Ages: 16 Years to 31 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Female participants
Study Population: This project will offer a PrEP delivery package within a prospective cohort study of sexually active HIV negative women ages 16-30 in locations in eSwatini, Kenya, Malawi, South Africa, Uganda, Zambia, and Zimbabwe to understand PrEP uptake, use, persistence and preferences for attributes of long-acting PrEP products and aspects of PrEP delivery for long-acting PrEP
Sampling Method: Probability Sample
Enrollment: 3087 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
A cohort for evaluation of open-label PrEP delivery and PrEP preferences among African women | 1 year
  We will collect data on STI prevalence, contraception use, sexual behavior, risk perception as correlates for PrEP uptake, persistence and adherence. Adherence will be measured by the timing of PrEP refills, self-reported PrEP use, and drug level testing for tenofovir (TFV) levels .PrEP adherence will be assessed during periods of risk, based on behavioral data and self-perceived risk. Participants in this cohort will be informed of other HIV prevention efficacy trials. A discrete choice experiment will be used to assess women's preferences around PrEP delivery form (pill and injection), dosing frequency, and relative dose forgiveness for different PrEP formulations. A patient-facing decision support tool about PrEP options will be evaluated with respect to its utility in assisting young women to consider their HIV prevention needs and PrEP preferences.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, Principal Investigator — University of Washington
Locations (20):
- ICAP, eSwatini Prevention Center, Mbabane, Hhohho Region, Eswatini
- Kenya Medical Research Institute (KEMRI), Nairobi, Kenya
- Queen Elizabeth Central Hospital, Blantyre, Malawi
- South Africa (14):
  - Perinatal HIV Research Unit (PHRU), Johannesburg, Gauteng
  - Wits Reproductive Health & HIV Institute (WRHI), Johannesburg, Gauteng
  - Helen Joseph Hospital--CHRU, Johannesburg, Gauteng
  - Human Sciences Research Council (HSRC), Pretoria, Gauteng
  - Setshaba Research Center, Pretoria, Gauteng
  - SA Medical Research Councit, Chatsworth, Chatsworth, KwaZulu-Natal
  - Maternal Adolescent & Child Health Research (MatCH), Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic, Ladysmith, KwaZulu-Natal
  - Madibeng Centre for Research, Brits, North West
  - Aurum Institute Klerksdorp (CRS), Klerksdorp, North West
  - Aurum Institute--Rustenburg, Rustenburg, North West
  - University of Cape Town--Khayekutsha, Cape Town, Western Cape
  - UCT-Masi, Cape Town, Western Cape
  - Emavundleni Research Center, DTHF, Nyanga, Western Cape
- Makerere University, Kampala, Uganda
- Kamwala Health Centre, Lusaka, Lusake, Zambia
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mukui I, Peacock S, Donnell D, Gati-Mirembe B, Krows M, Bukusi EA, Imaan L, Kotze P, Gill KM, Macdonald P, Louw C, Jaggernath M, Marais A, Peters RPH, Delany-Moretlwe S, Ward A, du Preez P, Kasaro M, Gandhi M, Heffron R, Celum C; INSIGHT Study Team. High prevalence and incidence of curable sexually transmitted infections among young women using oral HIV pre-exposure prophylaxis in sub-Saharan Africa: results from the INSIGHT Cohort study. Sex Transm Infect. 2025 Dec 25:sextrans-2025-056625. doi: 10.1136/sextrans-2025-056625. Online ahead of print. PMID 41448908
- [Derived] Gati Mirembe B, Donnell D, Krows M, Zwane Z, Bukusi E, Panchia R, Louw C, Mwelase N, Selepe P, Senne M, Naidoo L, Chihana R, Kasaro M, Nuwagaba-Biribonwoha H, Kotze P, Gill K, MacDonald P, vanHeerden A, Bosman S, Jaggernath M, du Preez P, Ward A, Peters RPH, Delany-Moretlwe S, Peacock S, Johnson R, Caucutt J, Morrison S, Wang G, Gandhi M, Velloza J, Heffron R, Celum C; INSIGHT Study Team. High recent PrEP adherence with point-of-care urine tenofovir testing and adherence counselling among young African women: results from the INSIGHT cohort. J Int AIDS Soc. 2024 Dec;27(12):e26389. doi: 10.1002/jia2.26389. PMID 39653676